CLINICAL TRIAL: NCT06343506
Title: Ankle Dorsiflexion Changes With Assisted Stretching Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Corey Alexander Pew, Assistant Professor, Montana State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-929-EXPEDITED
Record Dates: First submitted 2024-03-13; First posted 2024-04-02 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Physical Therapy Modality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Affected Individuals (Experimental)
  Interventions: Device: Grassroots Ankle Flex

INTERVENTIONS:
Device: Grassroots Ankle Flex — This device can be used in an individual's home, without assistance, allowing more frequent stretching without increased visits to physical therapy. The Ankle Flex device is used to stretch patients into a dorsiflexion position by securing the foot to the base of the device and the shin to the leg strap attached to the pulley system. The patients can then pull the handle of the pulley system, giving them the mechanical advantage to gently mobilize their ankle into dorsiflexion with their foot firmly secured to the base of the device. This can allow for a deeper and more controlled stretch than previous stretching methods done during at home care.

SUMMARY:
Ankle range of motion is an important degree of freedom for performing activities of daily living. Limited range of ankle motion has been related to Achilles tendonitis, lower limb injury, and abnormal gait leading to overuse injury. While stretching and massage can help increase range of motion the amount and frequency of manual manipulation needed to affect range of motion is not accessible to an individual in their home. A new device has been developed to allow deep stretching of the ankle and surrounding muscles to help increase ankle dorsiflexion. This device can be used in an individual's home, without assistance, allowing more frequent stretching without increased visits to physical therapy. The goal of this study is to determine the effect of using this device during a course of treatment to improve ankle dorsiflexion in individuals with decreased ankle range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of limited ankle range of dorsiflexion by physical therapist

Exclusion Criteria:

* Inability to perform testing activities as described in the consent form by self-report
* Inability to perform daily stretching with the device by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Ankle Range of Motion | Following 3 Weeks of Device Use
  Range of motion during passive and active movement.

SECONDARY OUTCOMES:
Ankle Strength | Following 3 Weeks of Device Use
  Strength in dorsiflexion

CONTACTS AND LOCATIONS:
Overall Officials: Corey Pew, PhD, Principal Investigator — Montana State University
Locations (1):
- Neuromuscular Biomechanics Laboratory, Bozeman, Montana, United States